CLINICAL TRIAL: NCT04843293
Title: The Effect of Breast Milk Smell on Early Feeding Cues, Transition Period to Oral Nutrition and Abdominal Perfusion in Preterm Newborns
Brief Title: The Effect of Breast Milk Smell on Nutrition in Preterms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Assoch Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUAdlt42
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Milk; Digestion; Nutrition; Smell Stimulation; Preterm Birth
Keywords: Breast Milk; Abdominal Perfusion; Preterm Newborn; Smell Stimulation; Feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: In this study, stratified sampling was used according to postmenstrual week (PW) and type of nutrition. In order to ensure homogeneity in the intervention and control groups, according to PW [28-(33+6)] and [34-35+6)], according to the type of nutrition [mixed nutrition (breast milk + formula milk)] and [breast milk] 4 layers were formed. Firstly, 56 preterm newborns were divided as random into intervention (group A) and control (group B). Groups A and B were stratified first to the PW, then according to the type of feeding. Permutation was also used to strike a balance between the strata. Block sets were generated for each combination of the prognostic factors (PW and type of nutrition). The intervention and control groups were then randomized into the strata using a random numbers table.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Olfactory stimulation group (Experimental): Preterm newborns in the initiative group were sniffed the smell of breast milk before and during feeding, except for routine application
  Interventions: Behavioral: Olfactory stimulation
- Control Group (No Intervention): Premature newborns in the control group feeds gavage according to the routine of the clinic, and no attempt will be made during feeding.

INTERVENTIONS:
Behavioral: Olfactory stimulation — Newborns in the experimental group will be given the smell of breast milk during 3 consecutive feedings and for 3 days in the morning. Smell stimulation will be started 1 minute before gavage feeding and the application of breast milk odor will continue until the feeding ends. A hand-cleaning researcher will drip 15 drops of breast milk on sterile gauze to apply the smell of breast milk. Sterile gauze dripped with breast milk will be placed as close to the newborn's nose as possible and not in contact with the newborn's skin. After the feeding of the newborn is completed, the application of the smell of breast milk will be terminated and the gauze will be removed from the incubator. A new sterile gauze will be used for each feeding, and these processes will be repeated with each smell stimulation for three days.
  Arms: Experimental Group: Olfactory stimulation group

SUMMARY:
The study was planned to determine the effect of breast milk odor applied during gavage feeding on early feeding cues of preterm newborns, the transition time to oral feeding and abdominal perfusion.

DETAILED DESCRIPTION:
It is known that nutrient odors stimulate the initiation of digestion. However, in preterm newborns who are fed by gavage or parenterally, exposure to the nutrient smell that initiates digestion disappears. For this reason, it is known that odor stimulation is applied to preterm newborns to improve nutrition. It is known that fragrances such as fragrant essential oils, the smell of breast milk, and amniotic fluid have positive effects such as shortening the transition time to oral feeding in preterm newborns, increasing nutritional tolerance and weight gain, increasing hunger symptoms, providing analgesic effect in painful procedures, and reducing hospital stay. However, no study was found to jointly evaluate the effect of odor stimulation with breast milk on early nutritional cues, transition time to oral nutrition and abdominal perfusion in preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* Born at 28-36 weeks of PW
* Birth weight >1000 gr
* 1. and 5. Apgar score average per minute ≥ 6
* Gavage method used in nutrition
* Intermittent infusion method used in nutrition,
* Not receiving mechanical ventilation / CPAP support,
* No medication or treatment is administered by the nasal route,
* Without nasal obstruction,
* Have not received any established medical diagnosis

Exclusion Criteria:

* Drugs that affect gastrointestinal function (drugs that facilitate gastric emptying and gastrointestinal passage of nutrients by increasing gastrointestinal tract motility, and drugs that reduce gastrointestinal tract motility)
* Newborns without breast milk
* Continuous infusion or parenteral feeding method is used in nutrition

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Newborn Information Form | First measurement, 5 minutes
  It is a form prepared by researchers in accordance with the literature (Yildiz ve ark. 2011, Pillai ve ark. 2018, Schriever ve ark. 2018, Neal-Kluever ve ark. 2019). In the form; gender of the baby, date of birth, method of birth, gestational week at birth, average apgar score (1. and 5. in minutes), birth weight, postnatal age, duration of transition to oral nutrition, daily body weight, nutrition frequency, amount of nutrition, food type, breast milk type, daily vomiting frequency and daily defecation frequency are information.
Abdominal Perfusion and Distension Follow-Up Form | Before 1 minute from feeding
  It is a form that contains information about abdominal perfusion level developed by researchers in accordance with the literature (Gay ve ark. 2011, Gillam-Krakauer ve ark. 2013, Thomas ve ark. 2018). Near Infrared Spectroscopy (NIRS) is a noninvasive device used in routine of neonatal intensive care unit and will be used in this study to determine the abdominal perfusion of the baby.
Early Feeding Tips Tracking Form | Before 1 minute from feeding
  The form developed by the researchers in line with the literature includes the physiological and behavioral hunger symptoms of the baby, which are accepted as criteria for starting oral feeding in babies and maintaining oral nutrition successfully and reliably (Kirk, Alder ve King 2007, Ludwig ve Waitzman 2007, White ve Parnell 2013, Holloway 2014, Lubbe 2018). The form consists of 9 items, and the answers to the items are in the form of Yes / No. Evaluation of the items in the form will be done simultaneously and separately by two observers (researcher and clinical nurse) right after the babies begin to feed, and interobserver agreement will be evaluated in order to test the reliability of the form.

SECONDARY OUTCOMES:
Abdominal Perfusion and Distension Follow-Up Form | The second measurement is 10, 30, 60 and 120 after feeding is completed. minutes.
  It is a form that contains information about abdominal perfusion level developed by researchers in accordance with the literature (Gay ve ark. 2011, Gillam-Krakauer ve ark. 2013, Thomas ve ark. 2018). Near Infrared Spectroscopy (NIRS) is a noninvasive device used in routine of neonatal intensive care unit and will be used in this study to determine the abdominal perfusion of the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, PhD, Principal Investigator — Selcuk University; Adalet Yucel, Master Student, Study Chair — Selcuk University; Hanifi Soylu, PhD, Study Director — Selcuk University
Locations (1):
- Sibel Kucukoglu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] Gay AN, Lazar DA, Stoll B, Naik-Mathuria B, Mushin OP, Rodriguez MA, Burrin DG, Olutoye OO. Near-infrared spectroscopy measurement of abdominal tissue oxygenation is a useful indicator of intestinal blood flow and necrotizing enterocolitis in premature piglets. J Pediatr Surg. 2011 Jun;46(6):1034-40. doi: 10.1016/j.jpedsurg.2011.03.025. PMID 21683194
- [Result] Gillam-Krakauer M, Cochran CM, Slaughter JC, Polavarapu S, McElroy SJ, Hernanz-Schulman M, Engelhardt B. Correlation of abdominal rSO2 with superior mesenteric artery velocities in preterm infants. J Perinatol. 2013 Aug;33(8):609-12. doi: 10.1038/jp.2013.3. Epub 2013 Feb 7. PMID 23392317
- [Result] Kirk AT, Alder SC, King JD. Cue-based oral feeding clinical pathway results in earlier attainment of full oral feeding in premature infants. J Perinatol. 2007 Sep;27(9):572-8. doi: 10.1038/sj.jp.7211791. Epub 2007 Jul 12. PMID 17625573
- [Result] Neal-Kluever A, Fisher J, Grylack L, Kakiuchi-Kiyota S, Halpern W. Physiology of the Neonatal Gastrointestinal System Relevant to the Disposition of Orally Administered Medications. Drug Metab Dispos. 2019 Mar;47(3):296-313. doi: 10.1124/dmd.118.084418. Epub 2018 Dec 19. PMID 30567878
- [Result] Pillai A, Albersheim S, Matheson J, Lalari V, Wei S, Innis SM, Elango R. Evaluation of A Concentrated Preterm Formula as a Liquid Human Milk Fortifier in Preterm Babies at Increased Risk of Feed Intolerance. Nutrients. 2018 Oct 4;10(10):1433. doi: 10.3390/nu10101433. PMID 30287775
- [Result] Thomas S, Nesargi S, Roshan P, Raju R, Mathew S, P S, Rao S. Gastric Residual Volumes Versus Abdominal Girth Measurement in Assessment of Feed Tolerance in Preterm Neonates: A Randomized Controlled Trial. Adv Neonatal Care. 2018 Aug;18(4):E13-E19. doi: 10.1097/ANC.0000000000000532. PMID 30015674
- [Result] Yildiz A, Arikan D, Gozum S, Tastekin A, Budancamanak I. The effect of the odor of breast milk on the time needed for transition from gavage to total oral feeding in preterm infants. J Nurs Scholarsh. 2011 Sep;43(3):265-73. doi: 10.1111/j.1547-5069.2011.01410.x. Epub 2011 Jul 25. PMID 21884372
- [Derived] Yucel A, Kucukoglu S, Soylu H. The Effect of Breast Milk Odor on Feeding Cues, Transition Time to Oral Feeding, and Abdominal Perfusion in Premature Newborns: A Randomised Controlled Trial. Biol Res Nurs. 2024 Jan;26(1):160-175. doi: 10.1177/10998004231200784. Epub 2023 Sep 8. PMID 37682253